CLINICAL TRIAL: NCT01904760
Title: The Effect of Dexmedetomidine on Agitation and Delirium in Patients After Free Flap Reconstructive Surgery
Brief Title: Dexmedetomidine to Prevent Agitation After Free Flap Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yang Xudong, vice director of the department of Anesthesiology, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PKUSSIRB-2012006
Record Dates: First submitted 2013-06-27; First posted 2013-07-22 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Agitation; Delirium
Keywords: agitation; delirium; dexmedetomidine; head and neck surgery; microvascular free tissue transfer; flap
MeSH Terms: conditions — Psychomotor Agitation; Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexmedetomidine (Experimental): Dexmedetomidine(4㎍/mL) : 0.5㎍/kg/hr infusion for 1 hour before operation is completed and 0.2-0.7㎍/kg/hr infusion continuously until 6:00am the next day.
  Interventions: Drug: Dexmedetomidine
- control (Placebo Comparator): Drug: Normal saline 0.9% (guess as 4㎍/mL) : 0.5㎍/kg/hr infusion for 1 hour before operation is completed and 0.2-0.7㎍/kg/hr infusion continuously until 6:00am the next day.
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine(4㎍/mL) : 0.5㎍/kg/hr infusion for 1 hour before operation is completed and 0.2-0.7㎍/kg/hr infusion continuously until 6:00am the next day.
  Other Names: Precedex
  Arms: dexmedetomidine
Drug: Saline placebo — Normal saline 0.9% (guess as 4㎍/mL) : 0.5㎍/kg/hr infusion for 1 hour before operation is completed and 0.2-0.7㎍/kg/hr infusion continuously until 6:00am the next day
  Arms: control

SUMMARY:
Reconstruction using microvascular free tissue flap has been an important management in patients with maxillofacial tumor. It is often characterised as long operation time, more traumatic and require restriction of patient's head movement postoperatively in order to prevent disruption of microvascular anastomosis. Agitation and delirium are common in patients with free flap surgery, which may lead to serious consequences such as self extubation, injury or even failure of the flap.

Dexmedetomidine is a sedative and co-analgesic drug with high specificity for α2-adrenoceptor. It is widely used in ICU sedation in general hospital. However its use after free flap surgery is not well documented. Furthermore the effect of Dexmedetomidine on preventing delirium has not been proved.

The investigators hypothesized that the use of Dexmedetomidine would reduce emergence agitation and prevent delirium in patients after free flap surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing selected maxillofacial surgery with free flap reconstruction
* American Society of Anesthesiologist(ASA) classification I and II

Exclusion Criteria:

* bradycardia (< 50 bpm)
* severe heart block
* low blood pressure(SBP<80mmHg)
* Known allergy to alpha 2 agonists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- School and Hospital of Stomatology, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine | Control
Started | 40 | 40
Completed | 39 | 40
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Control | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (15.0) | 50.6 (12.3) | 50.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 21 | 21 | 42
Region of Enrollment [Number; unit: participants]
  China | 39 | 40 | 79

OUTCOME MEASURES:

1. Primary Outcome: Agitation in PACU
Description: Patients are kept calm and cooperative in the PACU. Agitation is defined as Riker-Agitation Scale(SAS)>=5.
Time Frame: participants will be followed for the duration of PACU stay, an expected average of 12 hours
Measure: Number; unit: participants
Arm/Group | Dexmedetomidine | Control
Number analyzed (Participants) | 39 | 40
participants
  overall agitation in PACU | 15 | 18
  agitation after PACU admission | 4 | 12

2. Secondary Outcome: Postoperative Delirium
Description: Patients are sent back to wards the next morning after operation and followed up on each of the 5 days postoperatively. Delirium will be confirmed based on CAM-ICU method.
Time Frame: on each of the 5 days postoperatively
Measure: Number; unit: participants
Arm/Group | Dexmedetomidine | Control
Number analyzed (Participants) | 39 | 40
participants | 2 | 5

3. Other Pre Specified Outcome: Patients' Vital Signs in PACU
Description: Patient's vital signs including heart rate, blood pressure, pulse oxygen saturation and respiratory rate are monitored continuously in PACU and recorded on 1,2,4,6,12 hour after PACU admission.
Time Frame: participants will be followed for the duration of PACU stay, an expected average of 12 hours
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Use of Analgesics and Sedatives in PACU
Description: extra analgesics and sedatives will be given when patients are agitated or if the patients ask for them.
Time Frame: participants will be followed for the duration of PACU stay, an expected average of 12 hours
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Pain Score in PACU
Description: Patients' pain score are evaluated by a numerous scale(0-10) at 8am the next day, just before they leave PACU.
Time Frame: at 8 am the next day
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Sleep Quality in PACU
Description: Patients' sleep quality in PACU are evaluated by a numerous scale(0-10) at 8am the next day.
Time Frame: at 8am the next day
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Overall Feeling in PACU
Description: Patients' overall feeling in PACU are evaluated by a numerous scale(0-10) at 8am the next day.
Time Frame: at 8am the next day
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Sleep Quality Within 5 Days Postoperatively
Description: Participants are followed for 5 days after operation and their sleep quality are evaluated every afternoon on each of the 5 days.
Time Frame: on each of the 5 days postoperatively
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Pain Score Within 5 Days Postoperatively
Description: Participants are followed for 5 days after operation and their pain score are evaluated by VAS method every afternoon on each of the 5 days. Patients' pain score on maxillofacial region and flap donation region are evaluated respectively.
Time Frame: on each of the 5 days postoperatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine | Control
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 1/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dexmedetomidine (N=40) | Control (N=40)
hypotension in PACU (Vascular disorders) | 0/39 (0) | 1 (1)
bradycardia in PACU (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes